CLINICAL TRIAL: NCT07168395
Title: Pre-emptive RTO for An Early Detected Gastric Varices in CT/MR Angiogram Trial (PRADA Trial)
Brief Title: Pre-emptive RTO for An Early Detected Gastric Varices in CT/MR Angiogram Trial
Acronym: PRADA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Edward Wolfgang Lee, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-1721
Record Dates: First submitted 2025-09-01; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Gastric Varices
Keywords: varices; stomach; gastric; hepatic encephalopathy; gastric variceal bleeding; bleeding; retrograde transvenous obliteration
MeSH Terms: conditions — Esophageal and Gastric Varices; Varicose Veins; Hepatic Encephalopathy; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-selective beta blockers (Active Comparator): Non-selective beta blockers prescribed according to standard of care treatment guidelines. These may include propranolol, nadolol, and timolol.
  Interventions: Drug: Non-selective beta blockers
- Retrograde transvenous obliteration (RTO) (Active Comparator): Pre-emptive treatment with retrograde transvenous obliteration
  Interventions: Procedure: Retrograde transvenous obliteration

INTERVENTIONS:
Drug: Non-selective beta blockers — Non-selective beta blockers are used in patients who have not had a previous variceal bleed to prevent bleeding by reducing blood pressure in the liver. These drugs also work by blocking beta receptors that reduce cardiac output and by causing vessel constriction in the abdominal organs, which lowers blood flow to the liver and the existing varices.
  Arms: Non-selective beta blockers
Procedure: Retrograde transvenous obliteration — Pre-emptive retrograde transvenous obliteration will be performed in patients randomized to this arm to evaluate the effectiveness in decreasing gastric variceal bleeding. Either CARTO or PARTO (coil or plug-assisted retrograde transvenous obliteration) will be performed using EMBOLIZATION COILS or VASCULAR PLUGS of different sizes based on the size of the shunt. Additionally, Gelfoam (collagen sponges) slurry will be injected into the shunt and varices to completely obliterate them.
  Other Names: CARTO, PARTO, BRTO, RTO, RTOs
  Arms: Retrograde transvenous obliteration (RTO)

SUMMARY:
A number of treatment modalities are currently in use for gastric variceal bleeding (GVB). Balloon-occluded, plug-assisted, and coil-assisted retrograde transvenous obliteration (RTO) procedures are described in the literature as treatments for GVB after a bleeding episode occurs. Preliminary data suggests that prophylactic treatment of gastric varices may improve patient outcomes compared to conservative management. This study aims to compare pre-emptive treatment of gastric varices with current recommended medical management in a randomized prospective study design. Eligible patients will be randomized to receive RTO or to continue conservative management. Patients will be followed for up to 2 years for comparison of clinical outcomes, including episodes of gastric variceal bleeding, overall survival and transplant-free survival, complications, and secondary interventions.

DETAILED DESCRIPTION:
Gastroesophageal varices occur in approximately 50% of patients with liver cirrhosis. Specifically, gastric varices (GV) are responsible for roughly 10-30% of all variceal hemorrhage which is less than their counterpart esophageal varices. Despite their lower recurrence rates, gastric variceal bleeds (GVB) are associated with higher mortality, with an estimated 35-90% of patients developing rebleeding after achieving hemostasis.

Currently, there are several treatments for GVB that include endoscopic injection therapies, percutaneous antegrade transhepatic obliteration (ATO), transjugular portosystemic shunt placement (TIPS), splenic artery embolization (SAE), and surgical treatment. However, these procedures in previously studied trials have well-documented risks that compromise clinical outcomes. One specific interventional radiology procedure that has maintained a positive reputation in its use for gastric variceal bleeds is balloon-occluded retrograde transvenous obliteration (BRTO). This was first reported by Kanagawa et al. in the early 1990s; BRTO remains a well-accepted method of treatment of gastric fundal varices with gastrorenal or gastrophrenic shunts because of its minimally invasive nature and highly effective results, with studies showing up to 95% clinical success rate in stopping variceal bleeding. However, this procedure still has its own risks and limitations. For example, BRTO requires injection of a sclerosing agent (e.g. sodium tetradecyl sulfate or ethanolamine oleate), which has been associated with pulmonary venothrombotic embolization, portal vein thrombosis, anaphylactic reaction, hemolysis, renal tubular disturbance and acute renal failure. Furthermore, BRTO involves an indwelling occlusive balloon that remains inflated for hours, thus resulting in lengthy procedure times with increased necessary hospital resources and serious potential complication for balloon rupture. Despite these risks for BRTO complications, the procedure has been largely adopted by the IR community for its high success in controlling acute GVB, improving liver function, and well-documented improvement of hepatic encephalopathy.

In 2013, Gwon et al. modified BRTO with a vascular plug replacing the indwelling balloon to minimize the technical and clinical complications associated with BRTO with results suggesting plug-assisted RTO (PARTO) to be simple, safe, and an effective treatment for GV. A year later, Lee et al., presented their own preliminary findings with a modified BRTO procedure involving coils instead of balloons with the conclusion that coil-assisted retrograde transvenous obliteration (CARTO) treatment of portal hypertension variceal bleeding was a feasible and safer alternative than BRTO. A case report by Terada et al. highlighted the benefits to CARTO in a few ways: 1) if the shunt was not conducive to balloon placement then CARTO was a superior alternative 2) a steerable catheter reduced the required access routes and 3) steerable catheters allow for selective catheterization of acute-angle branching vessels. During the past decade, CARTO and PARTO have evolved as a simpler and possibly safer alternative to BRTO with comparable efficacy and favorable complication profiles. Yet, despite the promising preliminary results during these last decades on RTO for GVB, there is limited data in regard to its long-term efficacy. Furthermore, given the everchanging treatments for prophylactic treatment of GVB per AASLD guidelines, there is not enough data to support RTO as a preemptive intervention to protect against primary GVB. This study is aimed at exploring this latter question.

Per AASLD guidelines, primary prophylactic management for prevention of first GVB is a non-selective beta blocker. These same guidelines recommend against either TIPS or BRTO for primary prophylaxis of GVB. Yet the AASLD guidelines for treatment change considerably after patient endorses their first variceal bleeding. For instance, if the patient had a GOV1 hemorrhage, first-line treatment against gastric variceal rebleeding is both a non-selective beta blocker and an endoscopic variceal ligation. If the patient had a GOV2 or IGV1 hemorrhage, then first-line treatment against gastric variceal rebleeding can be either TIPS or BRTO. While these guidelines provide a framework for gastric variceal management, currently, non-selective beta-blockers serve as the only prophylactic treatment against primary GVB. The current study challenges this guideline to see whether CARTO or PARTO, a procedure with high efficacy and high safety profile, can be integrated as an alternative prophylactic treatment against primary GVB.

In the investigators' recent retrospective study (unpublished data), the investigators demonstrated that the cumulative survival rates in patients who received prophylactic CARTO/PARTO were 94% and 62% at 60 and 120 months. In contrast, those who received CARTO/PARTO for active bleeding were 43% and 0% at 60 and 120 months, respectively. There was a significant difference between the two groups (p=0.00035). This finding needs to be further investigated in prospective trials to validate these findings, which could potentially change how patients with GV are treated.

In this study, the investigators will perform a single-center, prospective, randomized controlled trial to evaluate the effectiveness in reducing primary GVB between preemptive RTO and the current conservative standard of care in patients with gastric varices. The results of this study will guide clinical practice and standard of care management of RTO as a possible alternative to prophylactic treatment against primary GVB. The study will also collect extensive follow-up care in all participants to continue cultivating data for RTO-associated complications and assessing its effect on necessary secondary interventions. As RTO procedures continue to evolve and become more widely used, this study will have the ability to contribute important information towards the indication and guidance of CARTO as an alternative prophylactic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Patients with compensated cirrhosis with a higher risk of decompensation based on AASLD 2023 Practice Guidance (Kaplan et al) - no ascites with endoscopic visualization of varices
3. Confirmed diagnosis of gastric varices either through CT, MRI, or Endoscopy.
4. No imaging (LIRAD4 or 5) or tumor marker (AFP) evidence of HCC or other malignancy
5. MELD < 20
6. First de novo RTO procedure
7. Taking NSBB
8. Patent internal jugular or right common femoral vein
9. Willing to provide the hepatology service information for F/U
10. No known diagnosis of hypercoagulopathy
11. Patent portal vein or portal vein cavernous transformation

Exclusion Criteria:

1. Age <18 years
2. Patients with decompensated cirrhosis based on AASLD 2023 Practice Guidance (Kaplan et al)
3. Cardiac failure
4. Active variceal bleeding
5. History of gastroesophageal variceal bleeding
6. Previous TIPS, BRTO, CARTO or PARTO procedure
7. No right jugular or right common femoral venous access
8. No portal vein flow
9. Malignancy
10. Life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Episodes of variceal bleeding | 2 years
  To monitor and assess the effectiveness of decreasing gastric variceal bleeding episodes between those receiving pre-emptive retrograde transvenous obliteration versus conservative management with non-selective beta blockers.

SECONDARY OUTCOMES:
Complications | 2 years
  To compare complications related to retrograde transvenous obliteration versus conservative management with non-selective beta blockers, including worsening of gastric varices, other bleeding, ascites, or hepatic encephalopathy
Transplant-free survival | Two years
  To compare the short term (1 month), mid-term (3 months and 6 months), and long-term (every 3 months up to two years) outcomes of episodes of gastric variceal bleeding, overall survival and transplant-free survival, complications, and secondary interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Edward W. Lee, MD, PhD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Terada K, Ogi T, Yoneda N, Yokka A, Sugiura T, Koda W, Kobayashi S, Gabata T. Coil-assisted retrograde transvenous obliteration (CARTO) for the treatment of gastric varices via a single access route using steerable microcatheter: a case report. CVIR Endovasc. 2020 Jun 14;3(1):30. doi: 10.1186/s42155-020-00124-3. PMID 32537683
- [Background] Gwon DI, Ko GY, Yoon HK, Sung KB, Kim JH, Shin JH, Ko HK, Song HY. Gastric varices and hepatic encephalopathy: treatment with vascular plug and gelatin sponge-assisted retrograde transvenous obliteration--a primary report. Radiology. 2013 Jul;268(1):281-7. doi: 10.1148/radiol.13122102. Epub 2013 Mar 12. PMID 23481167
- [Background] Lee EW, Saab S, Gomes AS, Busuttil R, McWilliams J, Durazo F, Han SH, Goldstein L, Tafti BA, Moriarty J, Loh CT, Kee ST. Coil-Assisted Retrograde Transvenous Obliteration (CARTO) for the Treatment of Portal Hypertensive Variceal Bleeding: Preliminary Results. Clin Transl Gastroenterol. 2014 Oct 2;5(10):e61. doi: 10.1038/ctg.2014.12. PMID 25273155
- [Background] Miyoshi H, Ohshiba S, Matsumoto A, Takada K, Umegaki E, Hirata I. Haptoglobin prevents renal dysfunction associated with intravariceal infusion of ethanolamine oleate. Am J Gastroenterol. 1991 Nov;86(11):1638-41. PMID 1951242
- [Background] Hashizume M, Kitano S, Yamaga H, Sugimachi K. Haptoglobin to protect against renal damage from ethanolamine oleate sclerosant. Lancet. 1988 Aug 6;2(8606):340-1. doi: 10.1016/s0140-6736(88)92400-2. No abstract available. PMID 2899760
- [Background] Cho SK, Shin SW, Lee IH, Do YS, Choo SW, Park KB, Yoo BC. Balloon-occluded retrograde transvenous obliteration of gastric varices: outcomes and complications in 49 patients. AJR Am J Roentgenol. 2007 Dec;189(6):W365-72. doi: 10.2214/AJR.07.2266. PMID 18029851
- [Background] Kanagawa H, Mima S, Kouyama H, Gotoh K, Uchida T, Okuda K. Treatment of gastric fundal varices by balloon-occluded retrograde transvenous obliteration. J Gastroenterol Hepatol. 1996 Jan;11(1):51-8. doi: 10.1111/j.1440-1746.1996.tb00010.x. PMID 8672742
- [Background] Sarin SK, Lahoti D, Saxena SP, Murthy NS, Makwana UK. Prevalence, classification and natural history of gastric varices: a long-term follow-up study in 568 portal hypertension patients. Hepatology. 1992 Dec;16(6):1343-9. doi: 10.1002/hep.1840160607. PMID 1446890
- [Background] Wani ZA, Bhat RA, Bhadoria AS, Maiwall R, Choudhury A. Gastric varices: Classification, endoscopic and ultrasonographic management. J Res Med Sci. 2015 Dec;20(12):1200-7. doi: 10.4103/1735-1995.172990. PMID 26958057